CLINICAL TRIAL: NCT03465553
Title: Palliative Short Course Accelerated Radiation Therapy for Advanced Thoracic Cancer
Brief Title: Palliative Short Course Radiotherapy for Advanced Thoracic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARON LUNG
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Palliative Care
Keywords: palliative care; thoracic cancer; radiotherapy; pain; quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short course radiotherapy (Experimental): The radiotherapy is delivered over 2 days with accelerated hypo-fractionation.
  Interventions: Radiation: Short course radiotherapy

INTERVENTIONS:
Radiation: Short course radiotherapy — An accelerated hypo-fractionation radiotherapy is delivered for palliation in patients with advanced thoracic cancer

SUMMARY:
The study wants to define the maximum tolerated dose (MTD), safety and efficacy of a short course radiation therapy in patients with symptomatic advanced thoracic cancer.

DETAILED DESCRIPTION:
The study wants to define the maximum tolerated dose (MTD) of a conformal short course accelerated radiation therapy delivered in twice daily fractions and 2 consecutive days, and the feasibility of this fractionation in term of safety and efficacy for symptomatic palliation of advanced thoracic cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven advanced thoracic cancer
* excluded from curative therapy because of disease stage and/or presence of multiple comorbidities and/or poor performance status
* age > 18 years
* Eastern Cooperative Oncology Group (ECOG) <3

Exclusion Criteria:

- prior radiotherapy to the same region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  The maximum tolerated dose is defined as the dose level below the highest administered dose associated with dose limiting toxicity (DLT) in at least one third of patients

SECONDARY OUTCOMES:
Acute toxicity | 1 year
  Acute toxicity after treatment is evaluated with the Common Terminology Criteria for Adverse Events (CTCAE). Values range from 1 (minimum acute toxicity) to 5 (maximum acute toxicity).
Quality of life | 1 year
  Quality of life after the treatment is evaluated according with the Cancer Linear Analog Scale (CLAS). Values range from 0 (better status) to 10 (worst status).
Pain relief | 1 year
  Pain after treatment is evaluated with the Visual Analogic scale (VAS). Values range from 0 (no pain) to 10 (maximum possible pain).
Late toxicity | 1 year
  Late toxicity after the treatment is evaluated with the Toxicity criteria of the Radiation Therapy Oncology Group and the European Organization for Research and Treatment of Cancer (RTOG/EORTC). Values range from 1 (minimum late toxicity) to 5 (maximum/severe late toxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G. Morganti, MD, Principal Investigator — Radiation Oncology Center, Dept. of Experimental, Diagnostic and Specialty Medicine - DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, Italy
Locations (1):
- Radiation Oncology Center, Dept. of Experimental, Diagnostic and Specialty Medicine - DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farina E, Macchia G, Buwenge M, Siepe G, Zamagni A, Cammelli S, Cilla S, Wondemagegnhu T, Woldemariam AA, Uddin AFMK, Sumon MA, Cellini F, Deodato F, Morganti AG. Radiotherapy in palliation of thoracic tumors: a phase I-II study (SHARON project). Clin Exp Metastasis. 2018 Dec;35(8):739-746. doi: 10.1007/s10585-018-9942-6. Epub 2018 Oct 8. PMID 30298381